CLINICAL TRIAL: NCT04127578
Title: A Phase 1/2a Open-Label Ascending Dose Study to Evaluate the Safety and Effects of LY3884961 in Patients With Parkinson's Disease With at Least One GBA1 Mutation (PROPEL)
Brief Title: Phase 1/2a Clinical Trial of PR001 (LY3884961) in Patients With Parkinson's Disease With at Least One GBA1 Mutation (PROPEL)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Prevail Therapeutics (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: J3Z-MC-OJAA formerly PRV-PD101
Record Dates: First submitted 2019-10-14; First posted 2019-10-15 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Parkinson Disease
Keywords: Parkinson's Disease; GBA1 mutation; Glucocerebrosidase; PD-GBA; Parkinson's Disease Gene Therapy; AAV9; Gene Therapy; GBA; Gaucher Disease
MeSH Terms: conditions — Parkinson Disease; Gaucher Disease | interventions — Methylprednisolone; Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose Level 1 (Experimental)
  Interventions: Biological: LY3884961; Drug: Methylprednisolone; Drug: Sirolimus
- Dose Level 2 (Experimental)
  Interventions: Biological: LY3884961; Drug: Methylprednisolone; Drug: Sirolimus

INTERVENTIONS:
Biological: LY3884961 — Participants will receive a single dose of LY3884961, administered intra-cisterna magna
Drug: Methylprednisolone — 6 IV pulses administered as concomitant medication over 3 months
Drug: Sirolimus — Back-up treatment if corticosteroid is not well tolerated. Loading dose, followed by maintenance dose, followed by dose tapering; administered as concomitant medication

SUMMARY:
Study J3Z-MC-OJAA is a Phase 1/2a, multicenter, open-label, ascending dose, first in-human study that will evaluate the safety of intracisternal LY3884961 administration in patients with moderate to severe Parkinson's disease with at least 1 pathogenic GBA1 mutation. Two dose level cohorts of LY3884961 are planned (Dose Level 1 and Dose Level 2). The duration of the study is 5 years. During the first year, patients will be evaluated for the effect of LY3884961 on safety, tolerability, immunogenicity, biomarkers, and clinical efficacy measures. Patients will continue to be followed for an additional 4 years to continue to monitor safety as well as selected biomarker and efficacy measures.

ELIGIBILITY:
Inclusion Criteria:

* Body weight range of ≥40 kg (88 lbs) to ≤110 kg (242 lbs) and a body mass index (BMI) of 18 to 34 kg/m2.
* Diagnosis of Parkinson's Disease (PD) per UK Parkinson's Disease Society Brain Bank Clinical Diagnostic Criteria.
* Hoehn and Yahr Stage III-IV (as determined in Practically Defined OFF state).
* Stable use of background medications at least 8 weeks prior to investigational product (IP) administration, including but not limited to those used for treatment of PD. Gaucher Disease-PD patients receiving GD treatments should be on a stable regimen of their ERT or substrate replacement therapy (SRT) medication for at least 3 months prior to screening.
* At least 1 pathogenic GBA1 mutation confirmed by the central laboratory
* Negative screening test for Mycobacterium tuberculosis (MTB), documented negative MTB test within 1 year prior to Screening, or clearance by an infectious disease specialist.
* Patient and/or patient's legally authorized representative (LAR) has the ability to understand the purpose and risks of the study and provide written informed consent and authorization to use protected health information in accordance with national and local privacy regulations.
* Patient has a reliable study partner/informant (e.g., family member, friend) willing and able to participate in the study as a source of information on the patient's health status and cognitive and functional abilities (including providing input into the rating scales). The study partner should have regular contact with the patient (in person or via phone/video communication). The study partner must sign a separate partner informed consent form (ICF) indicating that she/he understands the study requirements and is willing to participate and attend study visits requiring study partner input.
* Women of nonchildbearing potential must be either surgically sterile or postmenopausal. Men and women of childbearing potential must use a highly effective method of contraception consistently and correctly for the duration of the study including the long-term follow-up. Individuals in an exclusively same sex relationship (as their preferred and usual lifestyle) are not required to use contraception.
* Men must agree to abstain from sperm donation for the duration of the study, including long-term follow-up.
* Women must agree to abstain from egg donation for the duration of the study, including long-term follow-up.
* Women of childbearing potential cannot be pregnant or lactating/breastfeeding and must have a negative result for serum pregnancy test at Screening.
* Patient is generally ambulatory, not dependent on walker or wheelchair
* Patient is living in the community (i.e., not in nursing home); some levels of assisted living may be permitted at the discretion of the Investigator.
* Pneumococcal and shingles vaccines are required within 10 years of Screening (allowed to be performed during Screening but must be given at least 4 weeks prior to start of the immunosuppressant treatment).
* Patient is up to date with age and gender-appropriate cancer screening as per local standard of care based on Principal Investigator's (PI) judgment.

Exclusion Criteria:

* Diagnosis of a significant CNS disease other than Parkinson's Disease (PD) that may be a cause for the patient's PD symptoms or may confound study objectives.
* MoCA (Montreal Cognitive Assessment) score of <14
* Spinal, cervical, or brain MRI/magnetic resonance angiography (MRA) indicating clinically significant abnormality, including evidence of prior hemorrhage, infarct >1 cm3 or >3 lacunar infarcts, or a structural abnormality deemed a contraindication to intracisternal injection.
* Hypersensitivity or contraindications to corticosteroid and/or, sirolimus use (including but not limited to osteoporosis with vertebral fractures within 1 year prior to Screening, uncontrolled hypertension, poorly controlled diabetes, uncontrolled hyperlipidemia or hypercholesterolemia as per Investigator assessment.
* Concomitant disease or condition within 6 months of Screening that could interfere with, or treatment of which might interfere with, the conduct of the study or that would, in the opinion of the Investigator, pose an unacceptable safety risk to the patient or interfere with the patient's ability to comply with study procedures; including, but not limited to the following:

  1. Evidence of clinically significant liver pathology;
  2. Unstable autoimmune disease; autoimmune disease requiring chronic immunosuppression;
  3. Poorly controlled/not adequately managed diabetes (Screening glycosylated hemoglobin [HbA1C] ≥ 7%);
  4. History of unstable angina, myocardial infarction, chronic heart failure (New York Heart Association Class III or IV), or clinically significant conduction abnormalities (e.g., unstable atrial fibrillation) within 1 year prior to Screening;
  5. Clinically significant 12-lead electrocardiogram (ECG) abnormalities at Screening, as determined by the Investigator;
  6. Uncontrolled hypertension;
  7. History of cancer, including B-cell cancers, within 5 years of Screening with the exception of fully excised non-melanoma skin cancers, non-metastatic prostate cancer, and full treated ductal carcinoma in situ, provided it has been stable for at least 6 months;
  8. History or current alcohol or drug abuse within 2 years of Screening;
  9. Any current psychiatric diagnosis that may interfere with patient's ability to perform study procedures and all assessments;
  10. At imminent risk of self-harm;
  11. Any medical disorders that, in the opinion of the Investigator, could interfere with study-related procedures (including safe performance of lumbar puncture [LP] or intracisternal injection), such as prohibitive spinal diseases, bleeding diathesis, clinically significant coagulopathy,, thrombocytopenia, or increased intracranial pressure;
  12. Documented stroke or transient ischemic attack within 1 year prior to Screening;
  13. History of seizure or unexplained blackouts within 10 years prior to Screening;
  14. Currently active infection or a severe infection (e.g., pneumonia, septicemia, central nervous system infections [e.g. meningitis, encephalitis]) within 12 weeks prior to Screening;
  15. History of severe allergic or anaphylactic reactions. History of hypersensitivity to any inactive ingredient of the IP or protocol-required immunosuppressant medications.
  16. Acute or chronic: hepatitis B (HBV); hepatitis C (HCV) infection must have completed curative antiviral treatment with HCV viral load below the limit of quantification or be HCV RNA negative due to prior treatment or natural resolution to be eligible for enrollment.
* Clinically significant abnormalities in laboratory test results at Screening.
* Participation within 3 months prior to Screening in another therapeutic investigational drug or device study with purported disease-modifying effects on PD, unless it can be documented that the patient received placebo.
* History of deep brain stimulator placement, focused ultrasound, or surgery for PD
* Any type of prior gene or cell therapy.
* Immunizations (live vaccines) in the 4 weeks prior to Screening. Note: Pneumococcal and shingles vaccine administrations are allowed during the Screening period (patients not previously vaccinated should receive pneumococcal and/or shingles vaccine administration at least 4 weeks prior to initiation of Immunosuppression regimen).
* Use of ambroxol within 8 weeks of dosing.
* Use of blood thinners in the 2 weeks prior to Screening lumbar puncture (LP) or intra-cisterna magna (ICM) procedure, or the anticipated need to initiate blood thinners during the study. Antiplatelet therapies (e.g., prophylactic aspirin, clopidogrel) are acceptable if the patient is medically able to temporarily stop 48 hours to 7 days (depending on the antiplatelet medication used) prior to and at least 48 hours after intracisternal injection and lumbar puncture.
* Contraindications or intolerance to imaging methods (MRI, MRA, CT, DaT-SPECT) inducing claustrophobia and/or intolerance to contrast agents used for MRI, MRA or CT.
* Contraindications to general anesthesia or deep sedation.
* Positive urine test for drugs of abuse (including opiates, benzodiazepines, amphetamines, cocaine, barbiturates, and phencyclidine) without prescription, at Screening and Day -1. Note: Use of medical marijuana is permitted provided the patient is on a stable regimen. It is also permitted if the patient resides in a state in which the recreational use of marijuana is legalized, so long as the patient does not meet drug abuse criteria (as defined in the Diagnostic and Statistical Manual of Mental Disorders Fifth Edition).
* Patient is generally frail or has any medical condition, for which, in view of the Investigator, participation in the study would not be in the best interest of the patient or is likely to prohibit further participation during the study.

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2020-01-03 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Cumulative number of Treatment-Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs) | 5 years
Incidence of procedure or treatment-emergent AEs measured by brain MRI, spine MRI and nerve conduction study (NCS) | 5 years
Treatment emergent immunogenicity of AAV9 in blood | Thru month 24
Change from baseline in immunogenicity of AAV9 in blood | Baseline and Month 24
Treatment emergent immunogenicity of GCase in blood | Thru Month 24
  GCase (glucocerebrosidase)
Change from baseline in immunogenicity of GCase in blood | Baseline and Months 24
  GCase (glucocerebrosidase)
Treatment emergent immunogenicity of Nfl in blood | Thru Month 24
  GCase (glucocerebrosidase)
Change from baseline in immunogenicity of Nfl in blood | Baseline and Month 24
  GCase (glucocerebrosidase)
Treatment emergent immunogenicity of AAV9 in CSF | Thru Month 24
Change in immunogenicity of AAV9 in CSF | Baseline and Month 12
Treatment emergent immunogenicity of GCase in CSF | Thru Month 24
Change in immunogenicity of GCase in CSF | Baseline, and Months 12

SECONDARY OUTCOMES:
Change in glycolipid levels in blood | Baseline, Days 7, 14, and 21, and Months 1, 1.5, 2, 3, 6, 9 and 12
Change in GCase levels | Baseline, Days 7, 14, and 21, and Months 1, 1.5, 2, 3, 6, 9 and 12
GCase enzyme activity levels in blood | Days 7, 14, and 21, and Months 1, 1.5, 2, 3, 6, 9 and 12
Change in glycolipid levels in CSF | Baseline, and Months 2, 6, and 12
Change in GCase levels in CSF | Baseline, and Months 2, 6, and 12
GCase enzyme activity levels in CSF | Months 2, 6, and 12

CONTACTS AND LOCATIONS:
Overall Officials: Travis B. Lewis, MD, PhD, Study Director — Prevail Therapeutics
Locations (15):
- United States (11):
  - Mayo Clinic, 13400 E. Shea Boulevard, Scottsdale, Arizona
  - Esperanza Clinical, 25220 Hancock Avenue, Murrieta, California
  - Rocky Mountain Clinical Research - CenExel - PPDS, 701 East Hampden Avenue Suite 510, Englewood, Colorado
  - K2 Medical Research, 101 Southhall Lane, Suite 150, Maitland, Florida
  - PPD, 100 West Gore Street, Suite 202, Orlando, Florida
  - Northwestern University Feinberg School of Medicine, Dept. of Neurology, Parkinson's Disease & Movement Disorders Center, 710 N. Lake Shore Drive, 11th Floor, Chicago, Illinois
  - Mayo Clinic, 200 First Street SW, Rochester, Minnesota
  - Mount Sinai Beth Israel, 10 Union Square East, Suite 5H, New York, New York
  - Joan and Sanford I. Weill Department of Medicine, 525 E 68th Street, New York, New York
  - Hospital of the University of Pennsylvania, 330 S. 9th Street, Philadelphia, Pennsylvania
  - Vanderbilt University Medical Center, 1500 21st Avenue South Suite 2600, Nashville, Tennessee
- Israel (4):
  - Shaare Zedek Medical Center, 12 Shmuel Biet Street, Jerusalem
  - Hadassah Medical Center, Hadassah Ein Kerem, Dept. of Neurology, P.O. Box 12000, Jerusalem
  - Sheba Medical Center, Tel Hashomer, Ramat Gan
  - Tel Aviv Sourasky Medical Center, 6 Weizmann St., Tel Aviv

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] De BP, Rosenberg JB, Selvan N, Wilson I, Yusufzai N, Greco A, Kaminsky SM, Heier LA, Ricart Arbona RJ, Miranda IC, Monette S, Nair A, Khanna R, Crystal RG, Sondhi D. Assessment of Safety and Biodistribution of AAVrh.10hCLN2 Following Intracisternal Administration in Nonhuman Primates for the Treatment of CLN2 Batten Disease. Hum Gene Ther. 2023 Sep;34(17-18):905-916. doi: 10.1089/hum.2023.067. PMID 37624739